CLINICAL TRIAL: NCT02152761
Title: A 24-week Double-blind Treatment and 24-week Follow-up, Randomized, Multicenter, Placebo-controlled, Phase IIa/IIb Study to Evaluate Safety and Efficacy of i.v. Bimagrumab on Total Lean Body Mass and Physical Performance in Patients After Surgical Treatment of Hip Fracture
Brief Title: Study of Efficacy and Safety of Bimagrumab in Patients After Hip Fracture Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBYM338D2201; 2013-003439-31 (EudraCT Number)
Record Dates: First submitted 2014-05-08; First posted 2014-06-02 (Estimated); Results first posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Muscle Wasting (Atrophy) After Hip Fracture Surgery
Keywords: bimagrumab; BYM338; hip fracture; elderly; controlled clinical trial; randomized; muscle wasting; atrophy
MeSH Terms: conditions — Muscular Atrophy; Atrophy; Hip Fractures | interventions — bimagrumab

STUDY DESIGN:
Intervention Model Description: randomized, interventional, multicenter, placebo-controlled, phase IIa/IIb trial in patients
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- bimagrumab 700 mg (Experimental): Approximately 70 patients who met all inclusion criteria and none of the exclusion criteria were treated with the bimagrumab high dose administered via intravenous infusion starting Day 1 until Week 20
  Interventions: Drug: bimagrumab
- bimagrumab 210 mg (Experimental): Approximately 70 patients who met all inclusion criteria and none of the exclusion criteria were treated with the bimagrumab medium dose administered via intravenous infusion starting Day 1 until Week 20
  Interventions: Drug: bimagrumab
- placebo (Placebo Comparator): Approximately 70 patients who met all inclusion criteria and none of the exclusion criteria received matching placbo administered via intravenous infusion starting Day 1 until Week 20
  Interventions: Other: placebo
- Bimagrumab 70 mg (Experimental): Approximately 35 patients who met all inclusion criteria and none of the exclusion criteria were treated with bimagrumad low dose administered via intravenous infusion starting Day 1 until Week 20
  Interventions: Drug: bimagrumab

INTERVENTIONS:
Drug: bimagrumab — Bimagrumab was administered as intravenous infusion starting on Day 1 until week 20.
  Other Names: BYM338
  Arms: Bimagrumab 70 mg; bimagrumab 210 mg; bimagrumab 700 mg
Other: placebo — Matching placebo was administered as intravenous infusion starting on Day 1 until week 20.
  Arms: placebo

SUMMARY:
The purpose of this study was to assess if bimagrumab is safe and effective in patients with muscle wasting (atrophy) after hip fracture surgery.

ELIGIBILITY:
Inclusion Criteria:

Must have X-ray confirmed successful hip fracture repair; Must have completed surgical wound healing; Ability to walk a specified distance with or without a walking aid; Must weigh at least 35 kg.

Exclusion Criteria:

Must not have history of any other lower limb fractures in the past 6 months; Must not have certain cardiovascular conditions; Must not have a chronic active infection (e.g. HIV, hepatitis B or C, etc); Must not have used high-dose corticosteroid medications for at least 3 months in the past year;

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2014-09-16 (Actual); Primary Completion 2018-05-14 (Actual); Study Completion 2018-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (50):
- United States (6):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, El Cajon, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Gainesville, Georgia
  - Novartis Investigative Site, Rochester, Minnesota
  - Novartis Investigative Site, New York, New York
- Novartis Investigative Site, Ciudad Autonoma de Bs As, Argentina
- Novartis Investigative Site, Bedford Park, South Australia, Australia
- Novartis Investigative Site, Graz, Austria
- Belgium (3):
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Ghent
- Novartis Investigative Site, Santiago, Chile
- Colombia (2):
  - Novartis Investigative Site, Cali, Valle del Cauca Department
  - Novartis Investigative Site, Barranquilla
- Czechia (6):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Hradec Králové, Czech Republic
  - Novartis Investigative Site, Pardubice, Czech Republic
  - Novartis Investigative Site, Pilsen, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Prague
- France (2):
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Montpellier
- Germany (4):
  - Novartis Investigative Site, Bad Abbach
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Würzburg
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Hatvan
- Japan (6):
  - Novartis Investigative Site, Nishinomiya, Hyōgo
  - Novartis Investigative Site, Kamakura, Kanagawa
  - Novartis Investigative Site, Kochi, Kochi
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Toyama, Toyama
- Mexico (2):
  - Novartis Investigative Site, Aguascalientes
  - Novartis Investigative Site, San Luis Potosí City
- Russia (3):
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Sestroretsk
  - Novartis Investigative Site, Yaroslavl
- Spain (3):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Geneva, Switzerland
- Taiwan (3):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
- Novartis Investigative Site, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Hofbauer LC, Witvrouw R, Varga Z, Shiota N, Cremer M, Tanko LB, Rooks D, Auberson LZ, Arkuszewski M, Fretault N, Schubert-Tennigkeit AA, Papanicolaou DA, Recknor C. Bimagrumab to improve recovery after hip fracture in older adults: a multicentre, double-blind, randomised, parallel-group, placebo-controlled, phase 2a/b trial. Lancet Healthy Longev. 2021 May;2(5):e263-e274. doi: 10.1016/S2666-7568(21)00084-2. PMID 36098133

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 384 subjects were screened, and 252 subjects completed Screening period. One was lost to follow-up after screening and did not attend any visits for treatment epoch therefore, 251 were recruited to study. 2 subjects died during Screening epoch (1 was reported as discontinued and 1 was reported as a screen failure)
Pre-assignment Details: 251 subjects entered treatment epoch and were randomized to one of the three bimagrumab dose groups (70 mg, 210 mg and 700 mg) or the placebo group. 1 from the 210 mg group was randomized in error and did not receive study drug. Of the 250 subjects who were randomized and treated, 207 completed the 24 weeks treatment epoch.
Groups:
- Bimagrumab 700 mg: bimagrumab 700mg administered via intravenous infusion from Day 1 until Week 20
- Bimagrumab 210 mg: bimagrumab 210 mg administered via intravenous infusion from Day 1 until Week 20
- Bimagrumab 70 mg: bimagrumad 70 mg administered via intravenous infusion starting Day 1 until Week 20
- Placebo: placbo administered via intravenous infusion from Day 1 until Week 20
Period: Epoch: Treatment Epoch
Arm/Group | Bimagrumab 700 mg | Bimagrumab 210 mg | Bimagrumab 70 mg | Placebo
Started | 75 | 70 | 34 | 72
Completed | 64 | 50 | 29 | 64
Not Completed | 11 | 20 | 5 | 8
Not completed — Technical problems | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 8 | 3 | 5
Not completed — Adverse Event | 3 | 6 | 1 | 2
Not completed — Death | 0 | 3 | 1 | 0
Not completed — Non-compliance with treatment | 1 | 1 | 0 | 0
Period: Epoch: Post-treatment Follow-up Epoch
Arm/Group | Bimagrumab 700 mg | Bimagrumab 210 mg | Bimagrumab 70 mg | Placebo
Started | 67 | 54 | 30 | 68
Completed | 63 | 47 | 30 | 66
Not Completed | 4 | 7 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 3 | 0 | 1
Not completed — Lost to Follow-up | 1 | 4 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) used for all efficacy analyses consists of all randomized patients who received at least one dose of treatment after randomization and had at least one post-dose efficacy assessment. Patients who were randomized in error were excluded. Patients were analyzed according to treatment they were assigned to at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimagrumab 700 mg | Bimagrumab 210 mg | Bimagrumab 70 mg | Placebo | Total
Number analyzed (Participants) | 75 | 69 | 34 | 72 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.1 (8.58) | 74.8 (8.94) | 76.1 (8.59) | 76.4 (7.88) | 75.8 (8.46)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 9 | 9 | 4 | 3 | 25
  65 - 74 years | 22 | 23 | 10 | 27 | 82
  75 - 84 years | 30 | 26 | 16 | 32 | 104
  =>85 years | 14 | 11 | 4 | 10 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 48 | 21 | 53 | 176
  Male | 21 | 21 | 13 | 19 | 74
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 57 | 58 | 26 | 53 | 194
  Black | 0 | 0 | 0 | 0 | 0
  Asian | 13 | 8 | 6 | 17 | 44
  Other | 4 | 3 | 2 | 2 | 11
  Native American | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Lean Body Mass Measured by DXA (Dual-energy X-ray Absorptiometry) at Weeks 12 and 24
Description: Mixed Model for Repeated Measures (MMRM) of change from baseline in total LBM (kg) by treatment and visit To assess dose-response relationship of bimagrumab and facilitate an adequate dose selection for future phase III studies, without the need for supportive data from another dose-response finding study, at least three doses were required, ranging from a non-effective or minimally effective dose to a dose where maximal efficacy is expected. Original study was initiated with only two doses of bimagrumab, therefore, a lower dose arm of 70mg has been added to this study with Amendment 2, changing the randomization ratio from 1:1:1 to 2:1:2:2 to either placebo, bimagrumab 70mg, bimagrumab 210mg, or bimagrumab 700mg. Since the 70mg dose was expected to show suboptimal efficacy and fewer patients were randomized to this group, it was used only for dose response modelling and not for hypothesis testing. Consequently, no efficacy evaluations for the bimagrumab 70mg Arm were performed
Time Frame: baseline, weeks 12 and 24
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: kg
Groups:
- Bimagrumab 700 mg; Bimagrumab 210 mg; Active Total Efficacy (AT:E): Change from baseline in total LBM
- Placebo: placebo
Arm/Group | Bimagrumab 700 mg | Bimagrumab 210 mg | Active Total Efficacy (AT:E) | Placebo
Number analyzed (Participants) | 75 | 69 | 144 | 72
kg
  week 12: number analyzed (Participants) | 62 | 52 | 114 | 66
  week 12 | 1.066 (0.0107) | 1.052 (0.0109) | 1.059 (0.0096) | 1.009 (0.0103)
  week 24: number analyzed (Participants) | 56 | 48 | 104 | 63
  week 24 | 1.064 (0.0113) | 1.042 (0.0115) | 1.053 (0.0101) | 0.996 (0.0109)
Statistical Analysis 1: Comparison: Bimagrumab 700 mg vs Placebo; week 12; Test type: Superiority; p < .0001, Mixed Models Analysis; Treatment Group Ratio (BYM - Placebo) = 1.057, 95% CI 2-sided [1.037 to 1.076] — Holm-Bonferroni method: Used to adjust the Type I error for two comparisons (BYM338 700 mg/Placebo) at Week 24. No control for multiplicity was made at Week 12
Statistical Analysis 2: Comparison: Bimagrumab 210 mg vs Placebo; week 12; Test type: Superiority; p < .0001, Mixed Models Analysis; Treatment group rratio (BYM - Placebo) = 1.043, 95% CI 2-sided [1.024 to 1.064] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Gait Speed at Week 24 (Meters/Sec)
Description: Mixed Model for Repeated Measures (MMRM) of change from baseline in derived gait speed (m/sec) by treatment and visit
  To assess dose-response relationship of bimagrumab and facilitate an adequate dose selection for future phase III studies, without the need for supportive data from another dose-response finding study, at least 3 doses were required, ranging from a non-effective or minimally effective dose to a dose where maximal efficacy is expected. Original study was initiated with only two doses of bimagrumab, therefore, a lower dose arm of 70mg was added to this study with Amendment 2, changing the randomization ratio from 1:1:1 to 2:1:2:2 to either placebo, bimagrumab 70mg, bimagrumab 210mg, or bimagrumab 700mg. Since the 70mg dose was expected to show suboptimal efficacy and fewer patients were randomized to this group, it was used only for dose response modelling and not for hypothesis testing. Consequently, no efficacy evaluations for the bimagrumab 70mg Arm were performed
Time Frame: Baseline, Week 24
Population: The Full Analysis Set (FAS) used for all efficacy analyses consisted of all randomized subjects who received at least 1 dose of investigational drug. Subjects were analyzed according to the treatment they were assigned to at randomization.
Measure: Least Squares Mean (Standard Error); unit: meters per second
Arm/Group | Bimagrumab 700 mg | Bimagrumab 210 mg | Placebo
Number analyzed (Participants) | 75 | 69 | 72
meters per second | 0.268 (0.0599) | 0.350 (0.0617) | 0.339 (0.0607)
Statistical Analysis 1: Comparison: Bimagrumab 700 mg vs Placebo; week 24; Test type: Superiority; p = 0.1829, Mixed Models Analysis — Treatment Difference (BYM-Placebo); LS Mean of Treatment Difference = -0.071, 95% CI 2-sided [-0.175 to 0.034]
Statistical Analysis 2: Comparison: Bimagrumab 210 mg vs Placebo; week 24; Test type: Superiority; p = 0.8365, Mixed Models Analysis; LS Mean of Treatment Difference = 0.011, 95% CI 2-sided [-0.096 to 0.119]

3. Secondary Outcome: Change From Baseline in Short Physical Performance Battery at Weeks 24
Description: MMRM change from baseline in total score by treatment & visit to Week 24 in physical performance measured by Short Physical Performance Battery (SPPB) that evaluates lower extremity function. Score range is 0 (worst performance) to 12 (best) to assess dose-response relationship of bimagrumab & facilitate adequate dose selection for future phase III studies, without need for supportive data from another dose-response finding study, at least 3 doses were required, ranging from non- or minimally effective dose to a dose where maximal efficacy was expected. Original study was initiated with only 2 doses, therefore, lower 70mg arm was added to this study, changing randomization ratio from 1:1:1 to 2:1:2:2 to either placebo, bimagrumab 70mg, 210mg, or 700mg. Since 70mg dose was expected to show suboptimal efficacy, fewer patients were randomized to this group & it was used only for dose response modelling & not hypothesis testing. Consequently, no efficacy evaluation for 70mg were performed
Time Frame: Week 24
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Bimagrumab 700 mg | Bimagrumab 210 mg | Placebo
Number analyzed (Participants) | 75 | 69 | 72
scores on a scale | 2.331 (0.5436) | 3.535 (0.5623) | 2.702 (0.5516)
Statistical Analysis 1: Comparison: Bimagrumab 700 mg vs Placebo; week 24; Test type: Superiority; p = 0.5802, Mixed Models Analysis; LS Mean of Treatment Difference = -0.371, 95% CI 2-sided [-1.311 to 1.053]
Statistical Analysis 2: Comparison: Bimagrumab 210 mg vs Placebo; week 24; Test type: Superiority; p = 0.0913, Mixed Models Analysis; LS Mean of the Treatment Difference = 0.833, 95% CI 2-sided [-0.135 to 1.801]

4. Secondary Outcome: Incidence of Falls up to Week 48
Description: Group falls rate
  The frequency of having at least one fall up to Week 48 was summarized by treatment groups
  Incidence of falls was calculated for each arm up to Week 48. The ratio of these fall rates versus Placebo were calculated and presented as the Falls Rate Ratio. As mentioned in comment 5.1 above, the Falls Rate Ratio for Placebo does not apply because it would entail comparing the group to itself
Time Frame: Up to Week 48
Population: The Full Analysis Set (FAS) used for all efficacy analyses consisted of all randomized subjects who received at least one dose of investigational drug. Subjects were analyzed according to the treatment they were assigned to at randomization
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of Falls per week
Groups:
- Bimagrumab 70mg: bimagrumab 70 mg administered via intravenous infusion from Day 1 until Week 20
Arm/Group | Bimagrumab 700 mg | Bimagrumab 210 mg | Bimagrumab 70mg | Placebo
Number analyzed (Participants) | 75 | 69 | 34 | 72
Number of Falls per week | 0.31 [0.14 to 0.70] | 0.45 [0.20 to 0.99] | 0.36 [0.13 to 0.97] | 0.29 [0.13 to 0.64]
Statistical Analysis 1: Comparison: Bimagrumab 700 mg vs Placebo; Test type: Superiority; p = 0.8353, Negative binomial regression; Falls Rate Ratio = 1.08, 95% CI 2-sided [0.53 to 2.21]
Statistical Analysis 2: Comparison: Bimagrumab 210 mg vs Placebo; Test type: Superiority; p = 0.2015, Negative binomial regression; Falls Rate Ratio = 1.58, 95% CI 2-sided [0.78 to 3.18]
Statistical Analysis 3: Comparison: Bimagrumab 70mg vs Placebo; week 24; Test type: Superiority; p = 0.3999, Negative binomial regression; Falls Rate Ratio = 1.25, 95% CI 2-sided [0.52 to 3.00]

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected for the maximum duration of treatment and follow up for a participant per protocol for approximately 48 weeks. All cause mortality (deaths) was collected from First Patient First Visit (FPFV) to Last Patient Last Visit (LPLV) up to a maximum of 48 weeks
Description: All cause mortality (on-treatment deaths) was collected for as long as participants could be contacted from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV) up to a maximum of 48 weeks
Groups:
- BYM338 700 mg: bimagrumab 700mg administered via intravenous infusion from Day 1 until Week 20
- BYM338 210 mg: bimagrumab 210mg administered via intravenous infusion from Day 1 until Week 20
- BYM338 70 mg: bimagrumab 70 mg via i.v. infusion
- AT:S: Active Total Safety
- Placebo: placebo administered via intravenous infusion from Day 1 until Week 20
Arm/Group | BYM338 700 mg | BYM338 210 mg | BYM338 70 mg | AT:S | Placebo
All-Cause Mortality (participants affected / at risk) | 1/75 | 3/69 | 1/34 | 5/178 | 1/72
Serious Adverse Events (participants affected / at risk) | 15/75 | 17/69 | 9/34 | 41/178 | 9/72
Other Adverse Events (participants affected / at risk) | 47/75 | 34/69 | 15/34 | 96/178 | 30/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BYM338 700 mg (N=75) | BYM338 210 mg (N=69) | BYM338 70 mg (N=34) | AT:S (N=178) | Placebo (N=72)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 1 | 3 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 1 | 3 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Enterobacter infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 2 | 1
Salpingo-oophoritis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Device breakage (Product Issues) | 0 | 0 | 0 | 0 | 1
Device dislocation (Product Issues) | 0 | 1 | 0 | 1 | 0
Device extrusion (Product Issues) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 3 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 1 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BYM338 700 mg (N=75) | BYM338 210 mg (N=69) | BYM338 70 mg (N=34) | AT:S (N=178) | Placebo (N=72)
Diarrhoea (Gastrointestinal disorders) | 7 | 4 | 0 | 11 | 1
Oedema peripheral (General disorders) | 9 | 3 | 1 | 13 | 4
Bronchitis (Infections and infestations) | 0 | 1 | 2 | 3 | 1
Nasopharyngitis (Infections and infestations) | 5 | 1 | 2 | 8 | 2
Urinary tract infection (Infections and infestations) | 8 | 3 | 2 | 13 | 2
Contusion (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 4 | 5
Fall (Injury, poisoning and procedural complications) | 14 | 12 | 6 | 32 | 13
Weight decreased (Investigations) | 4 | 4 | 1 | 9 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 6 | 5 | 19 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 1 | 10 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12 | 17 | 2 | 31 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 5 | 1
Cognitive disorder (Nervous system disorders) | 1 | 4 | 0 | 5 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 2 | 5 | 0
Hypertension (Vascular disorders) | 3 | 2 | 2 | 7 | 4

LIMITATIONS AND CAVEATS:
As there were no statistically significant improvements in functional measures (i.e. gait speed, SPPB) at week 24, the need to test for sustained improvement at wk 48 became irrelevant. So, wk 48 treatment differences were not evaluated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e.; data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT02152761/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/61/NCT02152761/SAP_001.pdf